CLINICAL TRIAL: NCT02432586
Title: Pilot Study: Intensive Education in a Residential Camp Setting for Families of Young Children With Type 1 Diabetes
Acronym: TotCamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 042014-061
Record Dates: First submitted 2015-03-10; First posted 2015-05-04 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM; Diabetes; Child; Toddler
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensive Education (Other): Attendance of 2 intensive education sessions
  Interventions: Behavioral: Intensive Education

INTERVENTIONS:
Behavioral: Intensive Education — Participants will attend a 3 day family-centered, multidisciplinary, intensive education session at our regional diabetes camp, Camp Sweeney. A second 'booster' session will be conducted 6 months later.

SUMMARY:
18 preschool aged children and their families will attend structured, multidisciplinary, family-centered intensive education sessions over a 3-day weekend in a residential camp setting to address the unique challenges of managing type 1 diabetes mellitus in young children. A second 'booster' session, will be conducted 6 months later.

DETAILED DESCRIPTION:
We propose to deliver a structured multidisciplinary family-centered intervention over a 3-day weekend, with a second similar "booster" session 6 months later. The intervention will be based at our regional diabetes camp, Camp Sweeney. The proposed camp encounters aim to provide:

* An opportunity for intensive education beyond that achievable in a single class, and without the unfavorable impacts of multiple weekday classes on family and work time.
* Varied educational modalities including didactic sessions, practical demonstrations and role playing.
* Close observation of each child throughout the day and night by experienced diabetes counselors and medical staff to identify and help correct maladaptive family behaviors.
* A safe environment where parents can participate in group therapy sessions without child care worries.
* An opportunity for age-appropriate child-centered educational and therapeutic activities.
* An opportunity for families to form mutually-supportive friendships.
* Fun weekends away where the parents have help caring for their diabetic children.

We will conduct this pilot study, which will enroll 18 preschool children age 3-5.5 years, with the goal of obtaining preliminary results for 15 subjects.

The primary outcome, to be determined approximately one month before and after each of the two camp sessions, is improvement in Hemoglobin A1c (HbA1c). This outcome will be compared with that of historical controls.

Exploratory Hypotheses:

Compared with pretreatment baseline and historical controls, subjects attending two 3-day sessions at a family diabetes camp will improve:

* HbA1c 3 months after the first camp session
* Hypoglycemia frequency, as measured by continuous glucose monitoring
* Medical system utilization, as measured by telephone call frequency and also by emergency room visits and hospitalizations
* Behavioral/QoL assessments, including the parents of young children version of the hypoglycemia fear survey (HFS-P-YC), the Behavioral Pediatrics Feeding Assessment Scale (BPFAS), and the general and diabetes modules of the PedsQL.
* Diabetes knowledge, assessed by questionnaire
* Development of friendships between subject families, assessed by questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age 3-5.5 years old (+/- 2 months) at the date of first camp session they are eligible to join.
* Child and Parents fluent in either English or Spanish.
* Type 1 diabetes mellitus diagnosed for at least 10 months previous to date of first camp they are eligible to join.
* Taking insulin
* Custodial parent or guardian (preferable both parents or guardians) willing to attend both session of camp and the activities scheduled for them.
* Parent or guardian must sign consent before any study procedures are performed.

Exclusion Criteria:

* Neonatal diabetes (diagnosis in the first 3 months of life) or documented MODY; i.e., a likely genetic form of diabetes rather than an autoimmune etiology.
* Post-surgical diabetes (e.g., pancreatectomy for congenital hyperinsulinism). Such patients often cannot secrete glucagon, leading to a particularly severe inability to defend against hypoglycemia.
* Other severe chronic disease (e.g., cancer, cystic fibrosis) which in the judgment of the investigator is likely to significantly affect glycemic control.
* Patients cannot be taking systemic corticosteroids at enrollment because of adverse effects on glycemic control, but we will not disqualify subjects who require such therapy during the study. Inhaled or topical corticosteroids are permissible.
* Patients with hypothyroidism or hyperthyroidism must be clinically euthyroid and have free T4 and TSH within age-appropriate reference ranges at last medically indicated testing. Patients with out of range values may be retested after medication dose adjustment.
* Developmental delay or behavioral disorder in the patient of sufficient severity, in the judgment of the investigator, to interfere with group activities.
* Medical or psychiatric disorder in a parent of sufficient severity, in the judgment of the investigator, to interfere with group activities.
* Celiac disease is not an exclusion criterion.

Ages: 34 Months to 68 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c one month pre-camp to one month post-camp Session 1 | One month pre-camp, one month post-camp
  As compared to historical controls
Change in Hemoglobin A1c one month pre-camp to one month post-camp Session 2 | One month pre-camp, one month post-camp
  As compared to historical controls

SECONDARY OUTCOMES:
Change in Hypoglycemia frequency one month pre-camp to one month post-camp Session 1 | One month pre-camp, one month post-camp
  As measured by continuous glucose monitoring, and quantitated as area under the curve for blood glucoses <70 mg/dL.
Change in Hypoglycemia frequency one month pre-camp to one month post-camp Session 2 | One month pre-camp, one month post-camp
  As measured by continuous glucose monitoring, and quantitated as area under the curve for blood glucoses <70 mg/dL.
Medical system utilization ( emergency room visits, hospitalizations related to T1DM) | Duration of participation in study, expected to be 10 months
  Composite measure. As compared to historical controls.
Change in PedsQL Family Impact Module one month pre-camp to one month post-camp Session 1 | One month pre-camp, one month post-camp
  Parent report
Change in PedsQL Family Impact Module one month pre-camp to one month post-camp Session 2 | One month pre-camp, one month post-camp
  Parent report
Change in PedsQL Pediatric Quality of Life Inventory one month pre-camp to one month post-camp Session 1 | One month pre-camp, one month post-camp
  Parent report for Toddlers, Parent report for Young Children, Young Child Report
Change in PedsQL Pediatric Quality of Life Inventory one month pre-camp to one month post-camp Session 2 | One month pre-camp, one month post-camp
  Parent report for Toddlers, Parent report for Young Children, Young Child Report
Change in PedsQL Diabetes Module one month pre-camp to one month post-camp Session 1 | One month pre-camp, one month post-camp
  Parent report for Toddlers, Parent report for Young Children, Young Child Report
Change in PedsQL Diabetes Module one month pre-camp to one month post-camp Session 2 | One month pre-camp, one month post-camp
  Parent report for Toddlers, Parent report for Young Children, Young Child Report
Change in Hypoglycemia Fear Survey one month pre-camp to one month post-camp Session 1 | One month pre-camp, one month post-camp
  Parents of young children version
Change in Hypoglycemia Fear Survey one month pre-camp to one month post-camp Session 2 | One month pre-camp, one month post-camp
  Parents of young children version
Change in Behavioral Pediatrics Feeding Assessment one month pre-camp to one month post-camp Session 1 | One month pre-camp, one month post-camp
  Behavior section
Change in Behavioral Pediatrics Feeding Assessment one month pre-camp to one month post-camp Session 2 | One month pre-camp, one month post-camp
  Behavior section

CONTACTS AND LOCATIONS:
Overall Officials: Perrin White, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No